CLINICAL TRIAL: NCT03045406
Title: Apixaban for the Treatment of Venous Thromboembolism in Patients With Cancer: A Prospective Randomized Open Blinded End-Point (Probe) Study
Brief Title: Apixaban for the Treatment of Venous Thromboembolism in Patients With Cancer
Acronym: CARAVAGGIO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fadoi Foundation, Italy (Other)
Collaborators: University Of Perugia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FADOI.03.2016
Record Dates: First submitted 2017-01-17; First posted 2017-02-07 (Estimated); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apixaban (Experimental): orally administered, at the dose of 10 mg bid for 7 days, followed by 5 mg bid (total period of treatment: six months)
  Interventions: Drug: Apixaban
- Dalteparin (Active Comparator): subcutaneously administered, at a dose of 200 IU/kg SC o.i.d for 1 month. Thereafter, dalteparin will be administered at a dose of 150 IU/kg o.i.d. for 5 months
  Interventions: Drug: Dalteparin

INTERVENTIONS:
Drug: Apixaban — Tablets
  Arms: Apixaban
Drug: Dalteparin — Injections
  Arms: Dalteparin

SUMMARY:
Apixaban for the treatment of venous thromboembolism in patients with cancer: a prospective randomized open blinded end-point (PROBE) study

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with a newly diagnosed, objectively confirmed: symptomatic or unsuspected, proximal lower-limb DVT or symptomatic PE or unsuspected PE in a segmental or more proximal pulmonary artery;
* Any type of cancer (other than basal-cell or squamous-cell carcinoma of the skin, primary brain tumor or intracerebral metastasis and acute leukemia);
* Signed and dated informed consent of the patient, available before the start of any specific trial procedure.

Exclusion Criteria:

* age <18 years;
* ECOG Performance Status III or IV;
* life expectancy of less than 6 months;

Related to anticoagulant treatment:

* administration of therapeutic doses of LMWH, fondaparinux, or unfractionated heparin (UFH) for more than 72 hours before randomization;
* 3 or more doses of a vitamin K antagonist before randomization;
* thrombectomy, vena cava filter insertion, or thrombolysis used to manage the index episode;
* indication for anticoagulant treatment for a disease other than the index VTE episode;

Related to bleeding risk:

* thienopyridine therapy (clopidogrel, prasugrel, or ticagrelor) or aspirin over 165 mg daily or dual antiplatelet therapy;
* active bleeding or a high risk of bleeding contraindicating anticoagulant treatment;
* recent (in the last 1 month prior to randomization) brain, spinal or ophthalmic surgery
* hemoglobin level lower than 8 g/dL (5.0 mmol/L) or platelet count <75x10^9/L or history of heparin induced thrombocytopenia;
* creatinine clearance < 30 ml /min based on the Cockcroft Gault equation;
* acute hepatitis, chronic active hepatitis, liver cirrhosis; or an alanine aminotransferase level 3 times or more and/or bilirubin level 2 times or more higher the upper limit of the normal range;
* uncontrolled hypertension (systolic BP> 180 mmHg or diastolic BP > 100 mmHg despite antihypertensive treatment);
* concomitant use of strong inhibitors or inducers of both cytochrome P-450 3A4 and P-Glycoprotein;

Standard criteria:

* bacterial endocarditis;
* hypersensitivity to the active substance or to any of the excipients of study drug;
* patients participation in other pharmaco therapeutic program with an experimental therapy that is known to effect the coagulation system;
* childbearing potential without proper contraceptive measures, pregnancy, or breast feeding;
* any condition that as judged by the Investigator would place the subject at increased risk of harm if he/she participated in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1170 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gualberto Gussoni, MD, Study Director — FADOI Foundation
Locations (127):
- United States (18):
  - University of Southern California, Los Angeles, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Brigham and Women's Hospital/DFCI, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - New York-Presbyterian Hospital, New York, New York
  - Staten Island University Hospital/Northwell Health, Staten Island, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Belgium (2):
  - Cliniques universitaires Saint-Luc, Brussels
  - KU Leuven, Leuven
- France (16):
  - Hôpital Privé Arras Les Bonnettes, Arras
  - CHU Bordeaux Hôpital Saint André, Bordeaux
  - Hopital Cavale Blanche, Brest
  - Hôpital des armées HIA Clermont Tonnerre, Brest
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Louis Mourier, Colombes
  - Centre Hospitalier Universitaire Dijon Bourgogne, Dijon
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - CH de Vendée Centre Hospitalier Départemental, La Roche-sur-Yon
  - Centre Hospitalier Emile Roux Le Puy-en-Velay, Le Puy-en-Velay
  - Université de Limoges, Limoges
  - Centre Hospitalier Universitaire Lyon-Sud, Lyon
  - Hopital Pasteur - Chu de Nice, Nice
  - Hôpital Europeen Georges Pompidou, Paris
  - Université Jean Monnet, Saint-Etienne
  - Hôpital Sainte Musse, Toulon
- Germany (5):
  - Klinikum Darmstadt, Darmstadt
  - Städtisches Klinikum Dresden-Friedrichstadt, Dresden
  - Universitäts GefäßCentrum (UGC), Dresden
  - Universitätskrankenhaus Hamburg-Eppendorf, Hamburg
  - Forschungszentrum Ruhr, Witten
- Israel (6):
  - Haemek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
- Italy (33):
  - AOU Ospedali Riuniti di Ancona, Ancona
  - AOSG Moscati, Avellino
  - Ospedale Sacro Cuore di Gesù Fatebenefratelli, Benevento
  - ASST Papa Giovanni XXIII, Bergamo
  - Ospedale Maggiore, Bologna
  - Ospedale San Giacomo Apostolo, Castelfranco Veneto
  - Ospedale di Cosenza, Cosenza
  - Ospedale SS Annunziata, Cuneo
  - AOU Careggi, Florence
  - AOU San Martino, Genova
  - AOU di Modena, Modena
  - AO di Rilievo Nazione Antonio Cardarelli, Napoli
  - Istituto Nazionale Tumori - IRCCS Fondazione Pascale, Napoli
  - Ospedale Buon Consiglio Fatebenefratelli, Napoli
  - Ospedale San Martino, Oristano
  - Azienda Ospedaliera di Padova, Padua
  - AO Ospedali Riuniti Villa Sofia, Palermo
  - Department of Internal Medicine - University of Perugia, Perugia
  - Ospedale SS Cosma e Damiano, Pescia
  - Ospedale di Piacenza, Piacenza
  - AOU Pisana, Pisa
  - Ospedale di Pitigliano, Pitigliano
  - Ospedale di Ravenna, Ravenna
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale San Giovanni Calibita Fatebenefratelli, Roma
  - Policlinico Agostino Gemelli, Roma
  - Ospedale S. Paolo, Savona
  - AO Santa Maria, Terni
  - Ospedale Cà Foncello, Treviso
  - Ospedale di Udine, Udine
  - AO Ospedale di Circolo e Fondazione Macchi, Varese
  - Ospedale Sacro Cuore-Don Calabria di Negrar-Verona., Verona
  - Ospedale San Bortolo, Vicenza
- Netherlands (12):
  - Ziekenhuisgroep Twente ZGT, Almelo
  - Academic Medical Centre, Amsterdam
  - Rijnstate Arnhem, Arnhem
  - Rode Kruis Ziekenhuis Beverwijk, Beverwijk
  - Amphia Hospital Breda, Breda
  - Slingeland Doetinchem, Doetinchem
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Medisch Spectrum Twente, Enschede
  - Leiden University Medical Center, Leiden
  - Erasmus MC, Rotterdam
  - Haaglanden Hospital Den Haag, The Hague
  - HagaZiekenhuis, The Hague
- Poland (6):
  - Szpital Brzozów, Brzozów
  - Świetokrzyskie Centrum Onkologii, Kielce
  - Opolskie Centrum Onkologii, Opole
  - Medical Centre for Postgraduate Education - ECZ-Otwock, Otwock
  - CMKP, Otwock
  - Wielkoposkie Centrum Onkologii, Poznan
- Portugal (3):
  - IPO Lisboa, Lisbon
  - IPO Porto, Porto
  - Tràs-Os Montes e Alto Douro, Vila Real
- Spain (21):
  - Hospital Torrecardenas, Almería
  - Hospital Sant Pau, Barcelona
  - Hospital Val d'Hebron, Barcelona
  - Sabadell Hospital, Barcelona
  - Fundación Jiménez Díaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Clara Campal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Fuenlabrada, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital La Paz, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital de Málaga, Málaga
  - Hospital Morales Meseguer, Murcia
  - Hospital Central de Asturias, Oviedo
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Marqués Valdecilla, Santander
  - Hospital Virgen del Rocio, Seville
  - Hospital Clínico Lozano Blesa, Zaragoza
- United Kingdom (5):
  - University Hospitals Bristol, Bristol
  - University Hospital of Wales, Cardiff
  - King's College Hospital, London
  - Royal Gwent Hospital, Newport
  - Oxford University Hospital, Oxford

REFERENCES:
- [Derived] Becattini C, Bauersachs R, Maraziti G, Bertoletti L, Cohen A, Connors JM, Manfellotto D, Sanchez A, Brenner B, Agnelli G. Renal function and clinical outcome of patients with cancer-associated venous thromboembolism randomized to receive apixaban or dalteparin. Results from the Caravaggio trial. Haematologica. 2022 Jul 1;107(7):1567-1576. doi: 10.3324/haematol.2021.279072. PMID 34382385
- [Derived] Giustozzi M, Connors JM, Ruperez Blanco AB, Szmit S, Falvo N, Cohen AT, Huisman M, Bauersachs R, Dentali F, Becattini C, Agnelli G. Clinical characteristics and outcomes of incidental venous thromboembolism in cancer patients: Insights from the Caravaggio study. J Thromb Haemost. 2021 Nov;19(11):2751-2759. doi: 10.1111/jth.15461. Epub 2021 Jul 29. PMID 34260816
- [Derived] Agnelli G, Becattini C, Meyer G, Munoz A, Huisman MV, Connors JM, Cohen A, Bauersachs R, Brenner B, Torbicki A, Sueiro MR, Lambert C, Gussoni G, Campanini M, Fontanella A, Vescovo G, Verso M; Caravaggio Investigators. Apixaban for the Treatment of Venous Thromboembolism Associated with Cancer. N Engl J Med. 2020 Apr 23;382(17):1599-1607. doi: 10.1056/NEJMoa1915103. Epub 2020 Mar 29. PMID 32223112

FDAAA 801 VIOLATIONS:
- Correction Confirmed — The responsible party has responded, and this matter was resolved administratively. — issued 2025-09-30, released 2025-06-20, posted 2026-01-19
- Violation Identified — The entry for this clinical trial was not complete at the time of submission, as required by law. This may or may not have any bearing on the accuracy of the information in the entry. — issued 2024-12-19, released 2019-11-13, posted 2025-01-08

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apixaban | Dalteparin
Started | 585 | 585
Completed | 399 | 382
Not Completed | 186 | 203

BASELINE CHARACTERISTICS:
Population: 9 and 6 patients for the Apixaban and Dalteparin group, respectively, did not received the assigned treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Dalteparin | Total
Number analyzed (Participants) | 576 | 579 | 1155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 199 | 210 | 409
  >=65 years | 377 | 369 | 746
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (11.3) | 67.2 (10.9) | 67.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 284 | 303 | 587
  Male | 292 | 276 | 568
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 456 | 469 | 925
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 107 | 99 | 206
Region of Enrollment [Number; unit: participants] — A total of 1,170 patients were enrolled. However, 9 in the Apixaban group and 6 in the Dalteparin group did not receive the assigned treatment. Thus, 1,155 patients received treatment (576 Apixaban, 579 Dalteparin), representing the Overall Number of Baseline Participants.
  participants
    Netherlands | 64 | 74 | 138
    Belgium | 2 | 7 | 9
    United States | 60 | 65 | 125
    Poland | 10 | 10 | 20
    Italy | 204 | 193 | 397
    United Kingdom | 14 | 18 | 32
    Israel | 18 | 8 | 26
    France | 102 | 90 | 192
    Portugal | 8 | 5 | 13
    Germany | 14 | 14 | 28
    Spain | 80 | 95 | 175

OUTCOME MEASURES:

1. Primary Outcome: Recurrent Venous Thromboembolism
Description: Primary efficacy outcome: objectively confirmed recurrent VTE occurring during the study period, that means the composite of:
  · proximal DVT of the lower limbs (symptomatic or unsuspected), DVT of the upper limb (symptomatic), PE (symptomatic or unsuspected)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Dalteparin
Number analyzed (Participants) | 576 | 579
Participants | 32 | 46

ADVERSE EVENTS:
Time Frame: 6 months treatment + 1 month follow-up
Description: No difference in definition
Arm/Group | Apixaban | Dalteparin
All-Cause Mortality (participants affected / at risk) | 135/576 | 153/579
Serious Adverse Events (participants affected / at risk) | 255/576 | 276/579
Other Adverse Events (participants affected / at risk) | 89/576 | 74/579
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=576) | Dalteparin (N=579)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (6) | 4 (4)
Anaemia Of Malignant Disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 2 (2)
Microcytic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anaemia Of Chronic Disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normocytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac Thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial Haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 2 (2)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 8 (10) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (8) | 9 (11)
Intestinal Obstruction (Gastrointestinal disorders) | 6 (6) | 4 (4)
Melaena (Gastrointestinal disorders) | 4 (4) | 2 (2)
Rectal Haemorrhage (Gastrointestinal disorders) | 4 (4) | 3 (3)
Ascites (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal Pseudo-Obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mesenteric Artery Thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombosis Mesenteric Vessel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diaphragmatic Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal Stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhagic Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Condition Aggravated (General disorders) | 22 (22) | 19 (24)
Pyrexia (General disorders) | 12 (13) | 9 (9)
Death (General disorders) | 11 (11) | 19 (19)
General Physical Health Deterioration (General disorders) | 4 (4) | 13 (13)
Fatigue (General disorders) | 2 (2) | 3 (3)
Pain (General disorders) | 2 (2) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 4 (4)
Hyperthermia (General disorders) | 1 (2) | 0 (0)
Malaise (General disorders) | 1 (2) | 2 (2)
Mucosal Inflammation (General disorders) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 1 (1) | 0 (0)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 2 (2)
Administration Site Haematoma (General disorders) | 0 (0) | 1 (1)
Generalised Oedema (General disorders) | 0 (0) | 1 (1)
Hyperthermia Malignant (General disorders) | 0 (0) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 2 (2) | 2 (2)
Portal Vein Thrombosis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder Perforation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 2 (2)
Pneumobilia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular Injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 12 (12) | 10 (11)
Sepsis (Infections and infestations) | 9 (9) | 11 (12)
Respiratory Tract Infection (Infections and infestations) | 5 (5) | 4 (5)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1)
Abdominal Abscess (Infections and infestations) | 2 (2) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2)
Lung Infection (Infections and infestations) | 2 (2) | 1 (1)
Abdominal Wall Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess Neck (Infections and infestations) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Infected Skin Ulcer (Infections and infestations) | 1 (1) | 0 (0)
Muscle Abscess (Infections and infestations) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic Abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Fungal (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 6 (8)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Biliary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device Related Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Listeriosis (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 5 (6) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 2 (2) | 2 (2)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 1 (1)
Anticoagulation Drug Level Above Therapeutic (Investigations) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 1 (1) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
General Physical Condition Abnormal (Investigations) | 0 (0) | 1 (1)
Troponin Increased (Investigations) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic Disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 69 (69) | 77 (77)
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases To Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases To Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 3 (3) | 2 (2)
Cerebral Artery Thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrospinal Fistula (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Nervous System Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neurological Decompensation (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal Nerve Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 8 (10) | 5 (5)
Renal Failure (Renal and urinary disorders) | 4 (4) | 6 (6)
Acute Kidney Injury (Renal and urinary disorders) | 3 (3) | 8 (9)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Prerenal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 15 (16)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 15 (16)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (8)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary Infarction (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchopleural Fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Laryngeal Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Artery Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Drug Reaction With Eosinophilia And Systemic Symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 4 (4) | 5 (5)
Elective Surgery (Surgical and medical procedures) | 2 (2) | 1 (1)
Cancer Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Colostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Ileostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Lung Lobectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Lung Neoplasm Surgery (Surgical and medical procedures) | 1 (2) | 0 (0)
Neurosurgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Vena Cava Filter Insertion (Surgical and medical procedures) | 0 (0) | 2 (2)
Autologous Bone Marrow Transplantation Therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Jejunostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Mastectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Pain Management (Surgical and medical procedures) | 0 (0) | 1 (1)
Vena Cava Filter Removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 5 (5) | 5 (5)
Haemorrhage (Vascular disorders) | 2 (2) | 1 (1)
Vena Cava Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Atheroembolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Artery Occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Artery Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Superior Vena Cava Syndrome (Vascular disorders) | 0 (0) | 1 (2)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=576) | Dalteparin (N=579)
Anaemia (Blood and lymphatic system disorders) | 33 (38) | 21 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 33 (38) | 24 (28)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 29 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT03045406/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT03045406/SAP_001.pdf
  • Informed Consent Form (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT03045406/ICF_002.pdf